CLINICAL TRIAL: NCT02004145
Title: Trial of a Positive Psychology Intervention to Reduce Suicide Risk in Patients With Major Depression
Brief Title: Trial of a Positive Psychology Intervention in Major Depressive Disorder
Acronym: HOPE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Collaborators: American Foundation for Suicide Prevention (Other)
Responsible Party: Principal Investigator, Jeff C. Huffman, MD, Medical Director, Blake 11, Massachusetts General Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2013P001234; SRG-2-019-12 (Other Grant/Funding Number: AFSP)
Record Dates: First submitted 2013-12-03; First posted 2013-12-06 (Estimated); Last update posted 2016-04-19 (Estimated); Status verified 2016-04

CONDITIONS: Major Depressive Disorder
Keywords: MDD; Positive Psychology; Suicidality
MeSH Terms: conditions — Depressive Disorder, Major; Suicidal Ideation | interventions — Psychology, Positive

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Positive Psychology (Experimental): The Positive Psychology intervention consists of 6 exercises that will be completed by the participant with the guidance of a trainer.
  Exercises:
  Gratitude for positive events
  Gratitude letter
  Performing acts of kindness
  Using personal strengths
  Enjoyable and meaningful activities:
  Repeating one of the previous exercises.
  Interventions: Behavioral: Positive Psychology
- Organizational Skills (Sham Comparator): The Control Condition consists of 6 exercises that will be completed by the participant with the guidance of a trainer.
  Exercises:
  Daily Events
  Health Events
  Morning and Evening Events
  Interactions with Others
  Leisure Time Activities
  Repeating one of the previous exercises.
  Interventions: Behavioral: Control Condition

INTERVENTIONS:
Behavioral: Positive Psychology — The Positive Psychology intervention consists of 6 exercises that will be completed by the participant with the guidance of a trainer.
  Arms: Positive Psychology
Behavioral: Control Condition — The Control Condition consists of 6 exercises that will be completed by the participant with the guidance of a trainer.
  Arms: Organizational Skills

SUMMARY:
In this study, the investigators will perform an exploratory randomized trial of Positive Psychology (PP). The trial will consist of 50 participants and will compare the impact of a phone-based PP intervention vs. an attentional control condition, in Major Depressive Disorder (MDD) patients who are hospitalized for SI or following a suicide attempt. This is a 12 week trial with 6 weeks of intervention and two blinded follow-up assessments at 6 and 12 weeks.

Specific Aim #1: To assess the feasibility and acceptability of the phone-based PP intervention in this high-risk population.

Hypotheses: The intervention will be feasible (with most patients completing at least 4/6 PP and with follow-up data from at least 80% of subjects). The ratings of ease and subjective helpfulness of the exercise and other mental states as measured before and after each PP exercise will be more than 6 out of 10 and higher than the same ratings obtained from subjects in the control condition.

Specific Aim #2: To examine the impact of the six-session PP intervention on positive psychological well-being.

Hypothesis: Compared to control subjects, subjects randomized to PP will have greater scores on scales of optimism (measured via the Life Orientation Test-Revised [LOT-R]), gratitude (Gratitude Questionnaire-6 [GQ-6]), and positive affect (Positive Affect Negative Affect Schedule [PANAS]) at 6 and 12 weeks.

Specific Aim #3 (primary aim): To assess the impact of the PP intervention on key suicide risk factors.

Hypothesis: PP subjects will have greater scores on scales of hopelessness (Beck Hopelessness Scale [BHS]; primary study outcome measure), suicidal ideation (SI) (Concise Health Risk Tracking scale [CHRT]), and depression (Quick Inventory of Depressive Symptomatology-Self Report [QIDS-SR]) at 6 and 12 weeks.

We will also measure impact on readmission and suicide attempts to assess these key outcomes.

DETAILED DESCRIPTION:
Participants will be randomized to receive the intervention or recollection (control) arm. They will be randomized by a random-number generator and will be assigned a condition after receiving baseline questionnaires. The RA/blinded assessor will be blind to the study condition. The interventionist and subjects will not be blind to the study condition.

Baseline assessments: After consent and eligibility rule outs, subjects will receive baseline questionnaires to assess hopelessness (BHS46), suicidality (CHRT47), depression (QIDS-SR48), and positive states (LOT-R,43 GQ-6,44 PANAS45). Then, subjects will be randomized via random number generator to receive the control or intervention condition.

After completing baseline questionnaires and receiving randomization, subjects in both groups will have a 20 minute initial in-hospital session ("week #1"), within a week of anticipated discharge, in which the interventionist will provide a treatment manual specific to their condition, review the rationale for the initial exercise, and assign the exercise. The next day, the exercise will be reviewed and an exercise assigned for the next week. Immediately after completing the exercise, subjects will rate (on a Likert scale of 1-5) ease of exercise completion, overall utility, and initial impact on hopelessness/optimism, to assess immediate effects.

After discharge from the hospital, subjects will have five 20 minute weekly phone sessions ("weeks #2-6") with a different exercise used each week (assigned in the same order to all subjects). The phone sessions will include: (a) review of the prior week's exercise (including subject ratings of ease and impact as in week #1), (b) discussion of the rationale and assignment of the next week's exercise via a guided review of the study manual, and (c) completion of the Clinical Status questions and the Clinical Global Improvement scale (CGI) to monitor symptoms and improvement. Sessions will be audiotaped and random sessions reviewed by our PP consultant to ensure fidelity to the intervention (and that other techniques, e.g., Cognitive Behavioral Therapy, are not used).

Positive psychology (intervention condition)

Exercises. These were selected based on their superior performance in our pre-pilot study and others' work:

* Gratitude for positive events: Subjects recall three events, small or large, in the preceding week that were associated with satisfaction, happiness, pride, or other positive states.
* Gratitude letter: Subjects write a letter of gratitude thanking a person for an act of kindness; subject may, at their discretion, share the letter with the other person.
* Performing acts of kindness: Subjects are instructed to complete three acts of kindness in one day. The acts can be small or large, planned or spontaneous, but must be expressly completed to be kind to another.
* Using personal strengths: Subjects undergo a brief assessment of personal strengths, then find a new way to use that strength in the next 24 hours.
* Enjoyable and meaningful activities: Subjects complete a series of self-selected activities that vary between those that bring immediate boosts in mood and those that are more deeply meaningful.
* Repetition of an exercise previously done.

Recollection (control condition) The recollection condition was selected because it has been used in a prior study by our team of a phone-based positive psychology intervention and it was found to be feasible and well-accepted. Each week, subjects will record recent life events in a manual without describing emotions associated with the events. The nature, setting, or type of events to be recorded will differ each week to provide variety and maintain subjects' interest. This will be described as an intervention that may assist with organization and hone recall of important life events. Also, as an attentional control, it has a parallel structure to the experimental arm with a treatment manual, weekly exercises, and weekly calls to review exercises.

Follow-up 6 and 12 week phone call. After completion of the intervention (6 weeks), and then at 12 weeks, a blinded study research assistant (RA) will call subjects at 6 and 12 weeks to repeat measures of hopelessness (BHS), suicidality (CHRT), depression (QIDS-SR) and positive states (e.g., GQ-6, PANAS, LOT-R). Subjects will also be asked to rate their overall satisfaction with the treatment they received for their cardiac condition (outside of this study) over the last 6 and 12 weeks on a scale of 1 (excellent) to 5 (poor). We will record specific times that subjects would prefer to be called (and not to be called) for future follow-ups, to reduce intrusion on subjects' lives. We will also send a postcard to subjects reminding them of their upcoming study phone call. The blinded assessor will make 2 follow-up phone calls (at 6 and 12 weeks) to gather information about outcomes. If subjects would rather complete the questions in written form rather than over the phone, we will send them a written packet at the time of each follow-up.

ELIGIBILITY:
Inclusion Criteria:

* Patient admitted to Massachusetts General Hospital inpatient psychiatric unit
* Age 18 and older
* Able to read/write in English
* SI documented on admission OR admission due to a suicide attempt
* Admission diagnosis of MDD (and current major depressive episode), confirmed using the Mini International Neuropsychiatric Interview (MINI) and inpatient chart review

Exclusion Criteria:

* Psychotic symptoms, as assessed using the MINI and inpatient chart review
* Cognitive disorder, assessed using a six-item cognitive screen developed for research
* Primary admission diagnosis of substance use disorder

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 65 (Actual)
Dates: Start 2013-10; Primary Completion 2015-09 (Actual); Study Completion 2015-09 (Actual)

PRIMARY OUTCOMES:
Change in BHS Scores | Baseline, 6 weeks, and 12 weeks
  The Beck Hopelessness Scale (BHS) is a validated, twenty item, self-report measure that assesses three major aspects of hopelessness: feelings about the future, loss of motivation, and expectations.

SECONDARY OUTCOMES:
Change in CHRT Scores | Baseline, 6 weeks, and 12 weeks
  The Concise Health Risk Tracking scale (CHRT) is a brief, twelve item, self-report and clinician rating of suicidal risk.
Change in QIDS-SR Scores | Baseline, 6 weeks, and 12 weeks
  The Quick Inventory of Depressive Symptomatology-Self Report (QIDS-SR) is a sixteen item, self-report measure of depressive symptom severity derived from the 30-item Inventory of Depressive Symptomatology (IDS).

OTHER OUTCOMES:
Change in LOT-R Scores | Baseline, 6 weeks, and 12 weeks
  The Life Orientation Test-Revised (LOT-R) is a validated, six item, self-report measure of optimism.
Change in GQ-6 Scores | Baseline, 6 weeks, and 12 weeks
  The Gratitude Questionnaire 6 is a brief, validated six-item measure of dispositional gratitude.
Change in PANAS Scores | Baseline, 6 weeks, and 12 weeks
  The Positive Affect Negative Affect Schedule (PANAS) consists of ten words that subjects rate on a 5-point likert scale to asses positive affect.
Ease of Exercises | Week 1, Week 2, Week 3, Week 4, Week 5, Week 6
  Ease of exercises will be measured by a self-report 10-point Likert scale (0=very difficult to complete, 10=very easy to complete). Ease will be defined as an average score of 6 or more on this scale.
Rate of Intervention Feasibility | 12 weeks
  Rate of intervention feasibility will be measured by the number of exercises and follow-up assessments completed by each subject. There are 6 exercises and 2 follow-up assessments in total . A good rate of completion will be defined as an average of 4 or more exercises completed and >80% of follow-up assessments completed per subject.
Immediate Impact of Exercises | Week 1, Week 2, Week 3, Week 4, Week 5, Week 6
  Immediate impact of exercises will be measured by three self-report 10-point Likert scales measuring hopelessness (0=not hopeless, 10=very hopeless), mental organization (0=not organized, 10=very organized), and optimism (0=not optimistic, 10=very optimistic). Immediate impact will be defined as an average score of 6 or more on these scales.
Readmissions | 12 weeks
  Number of readmissions to the hospital

CONTACTS AND LOCATIONS:
Overall Officials: Jeff C Huffman, MD, Principal Investigator — Massachusetts General Hospital
Locations (1):
- Massachusetts General Hospital, Boston, Massachusetts, United States

REFERENCES:
- [Derived] Witt KG, Hetrick SE, Rajaram G, Hazell P, Taylor Salisbury TL, Townsend E, Hawton K. Psychosocial interventions for self-harm in adults. Cochrane Database Syst Rev. 2021 Apr 22;4(4):CD013668. doi: 10.1002/14651858.CD013668.pub2. PMID 33884617